CLINICAL TRIAL: NCT01726517
Title: A Phase 2, Randomized, Open-Label Study of Sofosbuvir/GS-5885 Fixed-Dose Combination ± Ribavirin in Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Safety and Efficacy of LDV/SOF Fixed-Dose Combination (FDC) ± Ribavirin in HCV Genotype 1 Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0118
Record Dates: First submitted 2012-11-10; First posted 2012-11-15 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2014-11

CONDITIONS: Chronic Hepatitis C Virus
Keywords: HCV genotype 1 (GT-1); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; GS-5885; Ribavirin; Open Label; Sofosbuvir; Treatment-Naïve; Protease Inhibitors; PI
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- LDV/SOF 8 Weeks (TN) (Experimental): Treatment-naive (TN) participants will be randomized to receive LDV/SOF for 8 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 8 Weeks (TN) (Experimental): Treatment-naive participants will be randomized to receive LDV/SOF plus RBV for 8 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 12 Weeks (TN) (Experimental): Treatment-naive participants will be randomized to receive LDV/SOF for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF 12 Weeks (TE) (Experimental): Treatment-experienced (TE) participants (had virologic failure following prior therapy with a protease-inhibitor [PI]+pegylated interferon [PEG]+RBV regimen) will be randomized to receive LDV/SOF for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 12 Weeks (TE) (Experimental): Treatment-experienced participants (had virologic failure following prior therapy with a PI+PEG+RBV regimen) will be randomized to receive LDV/SOF plus RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV 90 mg/SOF 400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+RBV 12 Weeks (TE); LDV/SOF+RBV 8 Weeks (TN)

SUMMARY:
This study is to evaluate the safety, tolerability, and antiviral efficacy of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) with or without ribavirin (RBV), administered for 8 or 12 weeks of treatment in participants with chronic genotype 1 hepatitis C virus (HCV) infection who are treatment-naive, and for 12 weeks in participants who had previously received a regimen containing a protease inhibitor for the treatment of HCV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, with chronic genotype 1 HCV infection
* HCV RNA equal to or greater than 10,000 IU/mL at screening
* Cirrhosis determination; a liver biopsy may be required
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Current or prior history of clinical hepatic decompensation
* Hepatocellular carcinoma (HCC) or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Hyland, Study Director — Gilead Sciences
Locations (1):
- San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Lawitz E, Poordad FF, Pang PS, Hyland RH, Ding X, Mo H, Symonds WT, McHutchison JG, Membreno FE. Sofosbuvir and ledipasvir fixed-dose combination with and without ribavirin in treatment-naive and previously treated patients with genotype 1 hepatitis C virus infection (LONESTAR): an open-label, randomised, phase 2 trial. Lancet. 2014 Feb 8;383(9916):515-23. doi: 10.1016/S0140-6736(13)62121-2. Epub 2013 Nov 5. PMID 24209977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 22 October 2012. The last participant observation was on 13 January 2014.
Pre-assignment Details: 116 participants were screened.
Groups:
- LDV/SOF 8 Weeks (TN): Treatment-naive (TN) participants were randomized to receive ledipasvir (LDV) 90 mg/sofosbuvir (SOF) 400 mg for 8 weeks.
- LDV/SOF+RBV 8 Weeks (TN): Treatment-naive participants were randomized to receive LDV 90 mg/SOF 400 mg plus weight-based ribavirin (RBV) (1000-1200 mg) for 8 weeks.
- LDV/SOF 12 Weeks (TN): Treatment-naive participants were randomized to receive LDV 90 mg/SOF 400 mg for 12 weeks.
- LDV/SOF 12 Weeks (TE): Treatment-experienced (TE) participants (had virologic failure following prior therapy with a protease-inhibitor [PI]+pegylated interferon [PEG]+RBV regimen) were randomized to receive LDV 90 mg/SOF 400 mg for 12 weeks.
- LDV/SOF+RBV 12 Weeks (TE): Treatment-experienced participants (had virologic failure following prior therapy with a PI+PEG+RBV regimen) were randomized to receive LDV 90 mg/SOF 400 mg plus weight-based RBV (1000-1200 mg) for 12 weeks.
Period: Overall Study
Arm/Group | LDV/SOF 8 Weeks (TN) | LDV/SOF+RBV 8 Weeks (TN) | LDV/SOF 12 Weeks (TN) | LDV/SOF 12 Weeks (TE) | LDV/SOF+RBV 12 Weeks (TE)
Started | 20 | 21 | 19 | 19 | 21
Completed | 20 | 21 | 18 | 19 | 21
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants received at least 1 dose of study drug
Groups:
- LDV/SOF 8 Weeks (TN): Treatment-naive participants were randomized to receive LDV 90 mg/SOF 400 mg for 8 weeks.
- LDV/SOF+RBV 8 Weeks (TN): Treatment-naive participants were randomized to receive LDV 90 mg/SOF 400 mg plus weight-based RBV (1000-1200 mg) for 8 weeks.
- LDV/SOF 12 Weeks (TE): Treatment-experienced participants (had virologic failure following prior therapy with a PI+PEG+RBV regimen) were randomized to receive LDV 90 mg/SOF 400 mg for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 8 Weeks (TN) | LDV/SOF+RBV 8 Weeks (TN) | LDV/SOF 12 Weeks (TN) | LDV/SOF 12 Weeks (TE) | LDV/SOF+RBV 12 Weeks (TE) | Total
Number analyzed (Participants) | 20 | 21 | 19 | 19 | 21 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (10.7) | 50 (11.1) | 46 (11.6) | 54 (6.6) | 52 (9.8) | 50 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 8 | 4 | 7 | 34
  Male | 14 | 12 | 11 | 15 | 14 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 12 | 9 | 6 | 10 | 40
  Not Hispanic or Latino | 17 | 9 | 10 | 13 | 11 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 1 | 2 | 2 | 9
  White | 15 | 21 | 17 | 16 | 19 | 88
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis C Virus (HCV) Genotype [Number; unit: participants] — There are variations within HCV genotype 1 which are distinct enough to be referred to as genotypes 1a or 1b.
  participants
    1a | 17 | 19 | 17 | 18 | 16 | 87
    1b | 3 | 2 | 2 | 1 | 5 | 13
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 4 | 7 | 1 | 2 | 1 | 15
    CT | 12 | 11 | 14 | 13 | 11 | 61
    TT | 4 | 3 | 4 | 4 | 9 | 24
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.1 (0.82) | 6.0 (0.84) | 6.1 (0.79) | 6.3 (0.49) | 6.2 (0.42) | 6.1 (0.69)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 9 | 7 | 7 | 4 | 5 | 32
  ≥ 800,000 IU/mL | 11 | 14 | 12 | 15 | 16 | 68
Prior HCV Treatment and Response [Number; unit: participants] — Prior HCV treatment and response was only collected for treatment-experienced participants in the LDV/SOF 12 Weeks (TE) and LDV/SOF+RBV 12 Weeks (TE) groups.
  participants
    Non-responder to PI boceprevir | 0 | 0 | 0 | 9 | 9 | 18
    Relapse/Breakthrough to PI boceprevir | 0 | 0 | 0 | 2 | 2 | 4
    Non-responder to PI telaprevir | 0 | 0 | 0 | 3 | 6 | 9
    Relapse/Breakthrough to PI telaprevir | 0 | 0 | 0 | 5 | 4 | 9
Cirrhosis [Number; unit: participants]
  No | 20 | 21 | 19 | 8 | 10 | 78
  Yes | 0 | 0 | 0 | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Weeks (TN) | LDV/SOF+RBV 8 Weeks (TN) | LDV/SOF 12 Weeks (TN) | LDV/SOF 12 Weeks (TE) | LDV/SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 20 | 21 | 19 | 19 | 21
percentage of participants | 95.0 | 100.0 | 94.7 | 94.7 | 100.0

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The number of participants experiencing an adverse event leading to permanent discontinuation of study drug(s) was summarized.
Time Frame: Baseline to Week 12
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | LDV/SOF 8 Weeks (TN) | LDV/SOF+RBV 8 Weeks (TN) | LDV/SOF 12 Weeks (TN) | LDV/SOF 12 Weeks (TE) | LDV/SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 20 | 21 | 19 | 19 | 21
participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 2, 4, 8, and 24 Weeks After Discontinuation of Therapy (SVR2, SVR4, SVR8, and SVR24)
Description: SVR2, SVR4, SVR8, and SVR24 was defined as HCV RNA < LLOQ at 2, 4, 8, and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 2, 4, 8, and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Weeks (TN) | LDV/SOF+RBV 8 Weeks (TN) | LDV/SOF 12 Weeks (TN) | LDV/SOF 12 Weeks (TE) | LDV/SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 20 | 21 | 19 | 19 | 21
percentage of participants
  SVR2 | 100.0 | 100.0 | 100.0 | 94.7 | 100.0
  SVR4 | 100.0 | 100.0 | 100.0 | 94.7 | 100.0
  SVR8 | 95.0 | 100.0 | 100.0 | 94.7 | 100.0
  SVR24 | 95.0 | 100.0 | 94.7 | 94.7 | 100.0

4. Secondary Outcome: Percentage of Participants Experiencing Viral Breakthrough or Viral Relapse
Description: * Viral breakthrough was defined as HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment, confirmed with 2 consecutive values (second confirmation value could be posttreatment), or last available on-treatment measurement with no subsequent follow-up values.
  * Viral relapse was defined as HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement.
Time Frame: Baseline to Posttreatment Week 24
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 8 Weeks (TN) | LDV/SOF+RBV 8 Weeks (TN) | LDV/SOF 12 Weeks (TN) | LDV/SOF 12 Weeks (TE) | LDV/SOF+RBV 12 Weeks (TE)
Number analyzed (Participants) | 20 | 21 | 19 | 19 | 21
percentage of participants
  Viral breakthrough | 0 | 0 | 0 | 0 | 0
  Viral relapse | 5.0 | 0 | 0 | 5.3 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 12 plus 30 days
Arm/Group | LDV/SOF 8 Weeks (TN) | LDV/SOF+RBV 8 Weeks (TN) | LDV/SOF 12 Weeks (TN) | LDV/SOF 12 Weeks (TE) | LDV/SOF+RBV 12 Weeks (TE)
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/21 | 1/19 | 1/19 | 1/21
Other Adverse Events (participants affected / at risk) | 9/20 | 12/21 | 8/19 | 7/19 | 12/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 8 Weeks (TN) (N=20) | LDV/SOF+RBV 8 Weeks (TN) (N=21) | LDV/SOF 12 Weeks (TN) (N=19) | LDV/SOF 12 Weeks (TE) (N=19) | LDV/SOF+RBV 12 Weeks (TE) (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 8 Weeks (TN) (N=20) | LDV/SOF+RBV 8 Weeks (TN) (N=21) | LDV/SOF 12 Weeks (TN) (N=19) | LDV/SOF 12 Weeks (TE) (N=19) | LDV/SOF+RBV 12 Weeks (TE) (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 6
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 4
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 3 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years